CLINICAL TRIAL: NCT03898986
Title: The Effects of Attenuated Versus Inactivated Flu Vaccine in Twin Sets
Acronym: FLU-TW
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Philip Grant, Assistant Professor of Medicine (Infectious Diseases), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 50200; 5U19AI057229-15 (NIH)
Record Dates: First submitted 2019-03-30; First posted 2019-04-02 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MZ twins (IIV or LAIV4) (Experimental): Up to 20 healthy monozygotic (MZ) individual twin volunteers, 2-20 years old, will be randomized within the twin pair to receive either inactivated influenza vaccine quadrivalent (IIV4) Fluzone® Quadrivalent vaccine or live, attenuated influenza vaccine quadrivalent (LAIV4) FluMist® Quadrivalent. Each volunteer will complete a total of 3 visits: Day 0 (pre-immunization), Day 7 and Day 28 post-immunization. All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  Interventions: Biological: Live attenuated influenza vaccine (LAIV4); Biological: Inactivated Influenza Vaccine (IIV4)
- DZ twins (IIV or LAIV4) (Experimental): Up to 20 healthy dizygotic (DZ) individual twin volunteers, 2-20 years old, will be randomized within the twin pair to receive either inactivated influenza vaccine quadrivalent (IIV4) Fluzone® Quadrivalent vaccine or live, attenuated influenza vaccine quadrivalent (LAIV4) FluMist® Quadrivalent. Each volunteer will complete a total of 3 visits: Day 0 (pre-immunization), Day 7 and Day 28 post-immunization. All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  Interventions: Biological: Live attenuated influenza vaccine (LAIV4); Biological: Inactivated Influenza Vaccine (IIV4)

INTERVENTIONS:
Biological: Live attenuated influenza vaccine (LAIV4) — LAIV4 vaccine dosage is 0.2 mL. The vaccine will be administered as an intranasal spray. Each sprayer contains a single dose of FluMist® Quadrivalent; approximately one-half of the contents should be administered into each nostril. 0.1 mL (i.e., half of the dose from a single FluMist sprayer) is administered into each nostril while the recipient is in an upright position. Insert the tip of the sprayer just inside the nose and rapidly depress the plunger until the dose-divider clip stops the plunger. The dose-divider clip is removed from the sprayer to administer the second half of the dose (0.1 mL) into the other nostril.
  Other Names: FluMist® Quadrivalent
Biological: Inactivated Influenza Vaccine (IIV4) — IIV4 vaccine will be administered as a 0.5 mL dose, with a sterile, disposable syringe and needle by IM injection.
  Other Names: Fluzone® Quadrivalent vaccine

SUMMARY:
This is one project of a larger ongoing study related to the immune system's response to the flu virus. This study is designed to investigate the immune response to the live attenuated influenza vaccine (LAIV) vs. the Inactivated Influenza Vaccine (IIV) in identical and fraternal twins.

DETAILED DESCRIPTION:
This is a Phase I mechanistic study of licensed influenza vaccines. The study requires 10 monozygotic and 10 dizygotic sets of twins (40 total participants) to enroll.

The duration of the study for an individual volunteer will be 4 weeks including screening and active participation. The study has a total of 3 visits.

First visit: Procedures during this visit are: Informed consent process, enrollment, study assessments, 20 ml blood draw, and vaccination. Participants will be randomized to receive either LAIV or IIV.

The time required to complete the first study visit will be about 30-40 minutes.

2nd (day 7 post vaccination) and 3rd (day 28 post vaccination ) visit: 20 ml blood will be obtained and the visit will take approximately 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. 2-20 year old male and female patients
2. Willing and able to complete the informed consent process
3. Availability of twin pair also agreeable and eligible for study inclusion
4. Availability for follow-up for the planned duration of the study
5. Acceptable medical history by review of inclusion/exclusion criteria

Exclusion Criteria:

1. Prior off-study vaccination with seasonal influenza vaccine within three months of study vaccination
2. Life-threatening reactions to previous influenza vaccinations
3. Asthma (contraindication for receipt of LAIV4)
4. Allergy to egg or egg products or to vaccine components including gentamicin, gelatin, arginine or MSG.
5. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
6. History of immunodeficiency (including HIV infection)
7. Known or suspected impairment of immunologic function; may include significant liver disease, diabetes mellitus treated with insulin or moderate to severe renal disease
8. Hospitalization in the past year for congestive heart failure or emphysema.
9. Chronic Hepatitis B or C.
10. Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible). Use of oral steroids (<20mg prednisone-equivalent/day) may be acceptable after review by the investigator.
11. Participants in close contact with anyone who has a severely weakened immune system
12. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
13. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator might jeopardize volunteer safety or compliance with the protocol.
14. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
15. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. per day), Plavix, or Aggrenox will be reviewed by investigators to determine if study participation would affect the volunteer's safety or compliance with the protocol.
16. Has taken an influenza antiviral medication within 48 hours prior to study vaccination [If yes, may not eligible if unable to schedule at an appropriate interval].
17. Receipt of blood or blood products within the past 6 months or planned used during the study.
18. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
19. Receipt of an inactivated vaccine 14 days prior to study enrollment, or planned vaccinations prior to completion of last study visit (~ 14 days after study vaccination)
20. Receipt of a live, attenuated vaccine within 60 days prior to enrollment of planned vaccination prior to completion of last study visit (~ 14 days after study enrollment)
21. Need for allergy immunization (that cannot be postponed) until after the last study visit.
22. History of Guillain-Barre# syndrome
23. Pregnant woman
24. Breastfeeding woman
25. Use of investigational agents within 30 days prior to enrollment or planned use during the study.
26. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or donation of platelets within 2 weeks of enrollment or planned donation prior to completion of the last visit.
27. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Grant, Principal Investigator — Assistant Professor of Medicine (Infectious Diseases)
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Inactivated Influenza Vaccine (IIV): Participants were randomized to received IIV
- Live Attenuated Influenza Vaccine 4 (LAIV 4): The other twin set was randomized to the LAIV
Period: Overall Study
Arm/Group | Inactivated Influenza Vaccine (IIV) | Live Attenuated Influenza Vaccine 4 (LAIV 4)
Started | 9 | 9
Identical Twin | 2 | 2
Fraternal Twin | 7 | 7
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Live Attenuated Influenza Vaccine 4 (LAIV 4): The other twin set was randomized to the LAIV4
- Total: Total of all reporting groups
Arm/Group | Inactivated Influenza Vaccine (IIV) | Live Attenuated Influenza Vaccine 4 (LAIV 4) | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: HAI Titers
Description: Evaluate HAI titers in response to influenza vaccination. An HAI titer is a hemoglobin assay that correlates to protection from influenza infection; an HAI titer of 40 or greater is considered to be protective.
Time Frame: Day 28
Population: Data were not collected for this outcome measure.
Arm/Group | Inactivated Influenza Vaccine (IIV) | Live Attenuated Influenza Vaccine 4 (LAIV 4)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Inactivated Influenza Vaccine (IIV) | Live Attenuated Influenza Vaccine 4 (LAIV 4)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT03898986/Prot_000.pdf
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT03898986/ICF_001.pdf